CLINICAL TRIAL: NCT01049503
Title: Effect of pH and Fluoride Concentration of Liquid Dentifrices on Caries Control in a Fluoridated Area: a Randomized Clinical Trial
Brief Title: Effect of pH and Fluoride Concentration of Dentifrices on Caries Control
Acronym: EPHFCDCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marilia Afonso Rabelo Buzalaf, Chair professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: USP0162009
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Dental Fluorosis; Dental Caries
Keywords: Dentifrices; Fluoride; Nails; Plaque
MeSH Terms: conditions — Fluorosis, Dental; Dental Caries; Plaque, Amyloid | interventions — Dentifrices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Caries-active 550 ppm F, pH 7.0 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-active children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH
- Caries-active 550 ppm F, pH 4.5 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-active children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH
- Caries-active 1100 ppm F, pH 7.0 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-active children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH
- Caries-inactive 550 ppm F, pH 7.0 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-inactive children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH
- Caries-inactive 550 ppm F, pH 4.5 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-inactive children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH
- Caries-inactive 1100 ppm F, pH 7.0 (Active Comparator): This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration in the caries control of caries-inactive children of a fluoridated area. One drop of the LD (liquid dentifrice) should be used 3 times/day for 12 months.
  Interventions: Other: Low fluoride and conventional dentifrices with different pH

INTERVENTIONS:
Other: Low fluoride and conventional dentifrices with different pH — Comparison of different dentifrice fluoride concentrations and pH on caries control
  Other Names: Dentifrice with 550 ppm F (NaF) and neutral pH (7.0); Dentifrice with 550 ppm F (NaF) and acidic pH (4.5); Dentifrice with 1100 ppm F (NaF) and neutral pH (7.0)

SUMMARY:
This study aims to assess the overall effect of pH and fluoride concentration of liquid dentifrices in the control of children dental caries of a fluoridated area, through visual inspection and the quantitative light-induced fluorescence (QLF) method. Toenail F concentration of a subsample of the children enrolled will be evaluated, in order to assess F bioavailability from these formulations and the evaluation of the concentration of fluoride incorporated into the biofilm will be done 6 months after initiation of the dentifrices use.

DETAILED DESCRIPTION:
Dentifrices have been recognized as one of the contributors in the increased prevalence of dental fluorosis, due to the fact that children in early childhood usually eat lots of them during brushing. As an alternative to the reduction of fluorosis have been suggested to reduce the concentration of fluoride toothpaste, however, its efficacy is not well established, increasing when the pH of the toothpaste is acidic, with a greater diffusion of F in the enamel. Therefore, this study aims to assess the overall effect of pH and fluoride concentration of liquid dentifrices in the control of children dental caries of a fluoridated area. A randomized double-blind study will be conducted with approximately 360 children aged 2 to 4 years old at public daycare centers located in a fluoridated area. Children will be examined by two examiners and classified according to caries activity. For 12 months, children will use 3 times a day, one of the toothpaste to be tested, with different concentrations of fluoride and pH. At the end of this period, children will be examined by the same examiners to check the progression of lesions. Clinical examinations should be performed by 2 calibrated examiners (kappa 0.8) at baseline and after 12 months. The diagnostic criteria of caries activity (active, inactive) and integrity of the surface of the lesion will be used. There will be a quantitative assessment of carious lesions fluorescence with a portable QLF equipment. In half of the sample, nails and plaque will be collected 6 months after initiation of the dentifrices use. Samples of plaque will be analyzed for fluoride using an ion-specific electrode after diffusion with hexamethyldisiloxane-facilitated disiloxane (HMDS). The presence of nails F will be analyzed as described above. For statistical analysis will be used ANOVA and test for individual comparisons.

ELIGIBILITY:
Inclusion Criteria:

* >= 2 years and <= 4 years
* Not having participated in any other clinical study within 3 months prior to selection;
* Not having very large carious lesions or dentin sensitivity during the study (if this occurs, the child will be referred for treatment);
* Signature of informed consent by the parents

Exclusion Criteria:

* Using orthodontic appliances

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 315 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marília AR Buzalaf, PhD, Principal Investigator — Bauru Dental School, University of São Paulo
Locations (1):
- Public primary schools in Bauru, Bauru, São Paulo, Brazil

REFERENCES:
- [Derived] de Almeida Baldini Cardoso C, Mangueira DF, Olympio KP, Magalhaes AC, Rios D, Honorio HM, Vilhena FV, Sampaio FC, Buzalaf MA. The effect of pH and fluoride concentration of liquid dentifrices on caries progression. Clin Oral Investig. 2014 Apr;18(3):761-7. doi: 10.1007/s00784-013-1031-2. Epub 2013 Jul 20. PMID 23873319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double-blind clinical trial was approved by the Institutional Review Board of Bauru Dental School (protocol 016/2009). It involved 2 to 4-year-old children that attended five public primary schools, each localized in a different geographical region of Bauru, São Paulo, Brazil (0.6-0.8 ppm F in the drinking water).
Pre-assignment Details: From 876 children of the 5 selected schools, 487 did not fill the informed consent. From those who filled the informed consen, 74 missed the clinical examination day or filled the exclusion criteria (had participated in other researches in the last 3 months or children using orthodontic appliances). The total number of children enrolled was 315.
Groups:
- Caries-active 550 Ppm F, pH 7.0; Caries-active 550 Ppm F, pH 4.5; Caries-active 1100 Ppm F, pH 7.0: This arm aims to assess the overall effect of pH and fluoride concentration in the caries control of caries-active children of a fluoridated area
- Caries-inactive 550ppm F, pH 7.0; Caries-inactive 550 Ppm F, pH 4.5; Caries-inactive 1100 Ppm F, pH 7.0: This arm aims to assess the overall effect of pH and fluoride concentration in the caries control of caries-inactive children of a fluoridated area
Period: Overall Study
Arm/Group | Caries-active 550 Ppm F, pH 7.0 | Caries-active 550 Ppm F, pH 4.5 | Caries-active 1100 Ppm F, pH 7.0 | Caries-inactive 550ppm F, pH 7.0 | Caries-inactive 550 Ppm F, pH 4.5 | Caries-inactive 1100 Ppm F, pH 7.0
Started | 52 | 48 | 56 | 55 | 56 | 48
Completed | 41 | 36 | 32 | 29 | 29 | 40
Not Completed | 11 | 12 | 24 | 26 | 27 | 8
Not completed — Lost to Follow-up | 11 | 12 | 24 | 26 | 27 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Caries-active 550 Ppm F, pH 7.0 | Caries-active 550 Ppm F, pH 4.5 | Caries-active 1100 Ppm F, pH 7.0 | Caries-inactive 550ppm F, pH 7.0 | Caries-inactive 550 Ppm F, pH 4.5 | Caries-inactive 1100 Ppm F, pH 7.0 | Total
Number analyzed (Participants) | 52 | 48 | 56 | 55 | 56 | 48 | 315
Age, Customized [Number; unit: Participants]
  >= 2 years and <= 4 years | 52 | 48 | 56 | 55 | 56 | 48 | 315
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 32 | 30 | 27 | 24 | 167
  Male | 23 | 23 | 24 | 25 | 29 | 24 | 148

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Concentration of Fluoride Incorporated Into the Biofilm Done 6 Months After Initiation of Dentifrices Use.
Description: Samples of plaque were analyzed for fluoride using an ion-specific electrode after diffusion with hexamethyldisiloxane-facilitated disiloxane (HMDS).
Time Frame: 6 months
Population: The sample size was calculated according to Pessan et al. (2008). From the trial participants in the fluoridated area, a convenience sample of 47 children was randomly selected. They were randomly divided (block allocation) into 3 groups, according to the type of liquid dentifrice they had been using for 6 months.
Measure: Mean (Standard Deviation); unit: mmol/kg
Groups:
- 550 Ppm F, pH 7.0; 550 Ppm F, pH 4.5; 1100 ppmF , pH 7.0: This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration on the concentration of fluoride incorporated into the biofilm.
Arm/Group | 550 Ppm F, pH 7.0 | 550 Ppm F, pH 4.5 | 1100 ppmF , pH 7.0
Number analyzed (Participants) | 16 | 15 | 16
mmol/kg | 0.80 (0.08) | 1.32 (0.23) | 1.74 (0.24)
Statistical Analysis 1: Comparison: 550 Ppm F, pH 7.0 vs 550 Ppm F, pH 4.5 vs 1100 ppmF , pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov and Smirnov and Bartlett tests, respectively. Data were analyzed by 2-way RM-ANOVA after logarithmic transformation and Bonferroni's test; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Caries Progression in Caries-active Children After 1 Year, According to the Type of Dentifrice Used
Description: The lesions' progression or regression was evaluated by the data from the examinations at baseline and after 12 months. The net increment was calculated from the difference between lesions' progression and regression. The lesions were considered to have progressed when a sound surface or inactive noncavitated (INC) caries lesion was reevaluated after 12 months as an active noncavitated caries lesion (ANC) or cavity (untreated cavity or filled tooth). The lesions' regression was considered when an ANC lesion was reevaluated after 12 months as INC lesion or sound surface.
Time Frame: baseline and 12 months
Population: The sample size was based on a previous trial (Lima et al., 2008). Accordingly, 24 children per dentifrice treatment resulted in a 85% power (α=0.05) for detecting difference of 0.23 and 0.65 in caries increment in the caries-inactive and caries-active groups, respectively. All the children that remained in the study after 12 months were analyzed.
Measure: Mean (Standard Deviation); unit: progressed lesions/child
Arm/Group | Caries-active 550 Ppm F, pH 7.0 | Caries-active 550 Ppm F, pH 4.5 | Caries-active 1100 Ppm F, pH 7.0
Number analyzed (Participants) | 41 | 36 | 32
progressed lesions/child | 2.12 (3.85) | 0.97 (1.96) | 1.75 (2.78)
Statistical Analysis 1: Comparison: Caries-active 550 Ppm F, pH 7.0 vs Caries-active 550 Ppm F, pH 4.5 vs Caries-active 1100 Ppm F, pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov; Smirnov and Bartlett tests, respectively. Data from the clinical exams were evaluated by Kruskal-Wallis' test; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

3. Secondary Outcome: Caries Regression in Caries-active Children After 1 Year, According to the Type of Dentifrice Used
Description: as for outcome 2
Time Frame: baseline and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: regressed lesions/child
Groups:
- Caries-active 550ppmF, pH 7.0; Caries-active 550ppmF, pH 4.5; Caries-active 1100ppmF, pH 7.0: This arm aims to assess the overall effect of pH and fluoride concentration in the caries control of caries-active children of a fluoridated area
Arm/Group | Caries-active 550ppmF, pH 7.0 | Caries-active 550ppmF, pH 4.5 | Caries-active 1100ppmF, pH 7.0
Number analyzed (Participants) | 41 | 36 | 32
regressed lesions/child | 1.34 (1.24) | 1.44 (1.83) | 1.84 (1.57)
Statistical Analysis 1: Comparison: Caries-active 550ppmF, pH 7.0 vs Caries-active 550ppmF, pH 4.5 vs Caries-active 1100ppmF, pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov; Smirnov and Bartlett tests, respectively.Data from the clinical exams were evaluated by Kruskal-Wallis' test; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

4. Primary Outcome: Evaluation of the Concentration of Fluoride Incorporated Into Participants' Toenails 6 Months After Initiation of the Dentifrices Use.
Description: Samples of nails were analyzed for fluoride using an ion-specific electrode after diffusion with hexamethyldisiloxane-facilitated disiloxane (HMDS).
Time Frame: 6 months
Population: The sample size was calculated according to Buzalaf et al. (2009). From the trial participants in the fluoridated area, a convenience sample of 161 children was randomly selected. They were randomly divided (block allocation) into 3 groups, according to the type of liquid dentifrice they had been using for 6 months.
Measure: Mean (Standard Deviation); unit: µgF/g
Groups:
- 550 Ppm F, pH 7.0; 550 Ppm F, pH 4.5; 1100 Ppm F, pH 7.0: This arm aims to assess the overall effect of the dentifrice pH and fluoride concentration on the concentration of fluoride incorporated into the toenails.
Arm/Group | 550 Ppm F, pH 7.0 | 550 Ppm F, pH 4.5 | 1100 Ppm F, pH 7.0
Number analyzed (Participants) | 58 | 53 | 50
µgF/g | 1.73 (0.68) | 1.80 (0.92) | 2.56 (1.31)
Statistical Analysis 1: Comparison: 550 Ppm F, pH 7.0 vs 550 Ppm F, pH 4.5 vs 1100 Ppm F, pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov and Smirnov and Bartlett tests, respectively. Data were analyzed by One-way ANOVA after logarithmic transformation and Tukey's test; Test type: Superiority or Other; p < 0.05, ANOVA

5. Secondary Outcome: Caries Progression in Caries-active Children After 1 Year, According to the Type of Dentifrice Used Assessed by the Quantitative Light Induced Method (QLF)(Fluorescence Change (∆F in %))
Description: The white spot lesions' progression was also determined by the QLF in a subsample of 75 caries-active children. The images were captured from the deciduous teeth which had at least one smooth surface with a clinically visible ANC. For every lesion, the fluorescence change (∆F in %) and the area of the lesion (mm^2)(baseline - 12 months)were calculated by the software at the QLF threshold of 5%. A negative ∆F value indicates caries regression.
Time Frame: baseline and 12 months
Population: The sample size was calculated according to Tranaeus et al. (2001). All the children that remained in the study after 12 months were analysed.
Measure: Mean (Standard Deviation); unit: lesions/child
Arm/Group | Caries-active 550ppmF, pH 7.0 | Caries-active 550ppmF, pH 4.5 | Caries-active 1100ppmF, pH 7.0
Number analyzed (Participants) | 11 | 18 | 16
lesions/child | 2.66 (2.52) | -3.46 (5.65) | -2.72 (3.97)
Statistical Analysis 1: Comparison: Caries-active 550ppmF, pH 7.0 vs Caries-active 550ppmF, pH 4.5 vs Caries-active 1100ppmF, pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov; Smirnov and Bartlett tests, respectively. Data from fluorescence loss were evaluated by Kruskal-Wallis and Dunn's tests; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

6. Secondary Outcome: Caries Progression in Caries-active Children After 1 Year, According to the Type of Dentifrice Used Assessed by the the Quantitative Light Induced Method (QLF) (Lesion Area (mm^2))
Description: The white spot lesions' progression was also determined by the QLF in a subsample of 75 caries-active children. The images were captured from the deciduous teeth which had at least one smooth surface with a clinically visible ANC. For every lesion, the fluorescence change (∆F in %) and the area of the lesion (mm^2)(baseline - 12 months)were calculated by the software at the QLF threshold of 5%.
Time Frame: baseline and 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: lesions/child
Arm/Group | Caries-active 550ppmF, pH 7.0 | Caries-active 550ppmF, pH 4.5 | Caries-active 1100ppmF, pH 7.0
Number analyzed (Participants) | 11 | 18 | 16
lesions/child | -1.03 (1.22) | 0.13 (0.80) | -0.06 (0.80)
Statistical Analysis 1: Comparison: Caries-active 550ppmF, pH 7.0 vs Caries-active 550ppmF, pH 4.5 vs Caries-active 1100ppmF, pH 7.0; The softwares GraphPad InStat version 3.0 for Windows and GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov; Smirnov and Bartlett tests, respectively. Data from lesion area were evaluated by ANOVA after logarithmic transformation and Tukey's test; Test type: Superiority or Other; p < 0.05, ANOVA

7. Secondary Outcome: Caries Progression in Caries-inactive Children After 1 Year, According to the Type of Dentifrice Used
Description: The lesions' progression was evaluated by the data from the examinations at baseline and after 12 months. The lesions were considered to have progressed when a sound surface or inactive noncavitated (INC) caries lesion was reevaluated after 12 months as an ANC lesion or cavity (untreated cavity or filled tooth).
Time Frame: baseline and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: progressed lesions/child
Groups:
- Caries-inactive 550 Ppm F, pH 7.0; Caries-inactive 550 Ppm F, pH 4.5; Caries-inactive 1100 Ppm F, pH 7.0: This arm aims to assess the overall effect of pH and fluoride concentration in the caries control of caries-active children of a fluoridated area
Arm/Group | Caries-inactive 550 Ppm F, pH 7.0 | Caries-inactive 550 Ppm F, pH 4.5 | Caries-inactive 1100 Ppm F, pH 7.0
Number analyzed (Participants) | 29 | 29 | 40
progressed lesions/child | 0.14 (0.74) | 0.03 (0.18) | 0.10 (0.50)
Statistical Analysis 1: Comparison: Caries-inactive 550 Ppm F, pH 7.0 vs Caries-inactive 550 Ppm F, pH 4.5 vs Caries-inactive 1100 Ppm F, pH 7.0; GraphPad Prism version 4.0 for Windows (GraphPad Software, La Jolla, Ca, USA) were used. Data were checked for normality and homogeneity using Kolmogorov; Smirnov and Bartlett tests, respectively.Data from the clinical exams were evaluated by Kruskal-Wallis' test; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Caries-active 550 Ppm F, pH 7.0 | Caries-active 550 Ppm F, pH 4.5 | Caries-active 1100 Ppm F, pH 7.0 | Caries-inactive 550ppm F, pH 7.0 | Caries-inactive 550 Ppm F, pH 4.5 | Caries-inactive 1100 Ppm F, pH 7.0
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48 | 0/56 | 0/55 | 0/56 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48 | 0/56 | 0/55 | 0/56 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No